CLINICAL TRIAL: NCT04021667
Title: The Effect Of Indıvıdual And Group Breast Feedıng Traınıng Of Future Mother And Father At Postpartum Perıod On Breast Feedıng Self-Effıcacy And Attıtude:Randomızed Controlled Study
Brief Title: The Effect Of Indıvıdual and Group Breastfeedıng Traınıng Of Candidate Mother And Father
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, YEŞİM YEŞİL, Research Assistant, Ege University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 0000-0003-2847-6978
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Breastfeeding; Education
Keywords: Breastfeeding; Parents Training; Self-Effıcacy; Attitude
MeSH Terms: conditions — Breast Feeding; Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: The pregnant women and partners who came to the hospital were evaluated in terms of sample criteria and randomized sampling was divided into three groups.
  In order to be able to perform randomized sampling, the selection of the groups to the individual breastfeeding education, group breastfeeding education and control group was determined by throwing a coin.
  After the first group was identified, a research group was taken for each day.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INDIVIDUAL BREASTFEEDING TRAINING (Experimental): Individual Breastfeeding Training: Mother and father candidates who applied to the pregnant outpatient clinic and met the study criteria were included in the study.
  After the informed consent was signed, the socio-demographic questionnaire including obstetric history and breastfeeding history, IOWA infant nutrition attitude scale and Breastfeeding Self-Efficacy Scale were applied to the mother and father candidates.
  Interventions: Other: educational intervention
- GROUP BREASTFEEDING TRAINING (Experimental): Group Breastfeeding Training: Mother and father candidates who applied to the pregnant outpatient clinic and met the study criteria were included in the study.
  After the informed consent was signed, the socio-demographic questionnaire including obstetric history and breastfeeding history, IOWA infant nutrition attitude scale and Breastfeeding Self-Efficacy Scale were applied to the mother and father candidates.The groups were composed of five pairs of parents.
  Interventions: Other: educational intervention
- Control Group (No Intervention): Control Group: Mother and father candidates who applied to the pregnant outpatient clinic and met the study criteria were included in the study.After the informed consent was signed, the socio-demographic questionnaire including obstetric history and breastfeeding history, IOWA infant nutrition attitude scale and Breastfeeding Self-Efficacy Scale were applied to the mother and father candidates. Routine procedures were applied to the mother and father candidates.

INTERVENTIONS:
Other: educational intervention — İndividual and Group Breastfeeding Education:It was taken into consideration that mothers and fathers who do not have breastfeeding experience in the antenatal period feel better in terms of their perception of the education given, and education is provided with adult education principles.Breastfeeding training slides, cloth nipple model, dummy dolls were used during the training and lecture, demonstration and application and breastfeeding training were provided.At the end of the training, they were given time to ask questions and their feedback was received.Control Group:Routine procedures in the clinic were performed for the mother and father candidates.The data of the mother and father who came to the hospital for antenatal follow-up and control were collected in four stages.
  Arms: GROUP BREASTFEEDING TRAINING; INDIVIDUAL BREASTFEEDING TRAINING

SUMMARY:
Breast feeding is the primary step for healthy generations. Breast milk protects against diseases of childhood period starting from infancy till adulthood. Inspite of the benefits of breast milk due to various reasons a lot of women all around the world and in our country can not begin breast feeding and leave it at an early stage even if they start once. According to Turkey Population and Health Investigation (TPHI) data of 2013; while the rate of only breast feeding among; 0-1 month babies is 57.9%, among babies under 6 months this rate falls to 10.0%. In the case of maternals not carrying out the whole breast feeding conditions situations such as milk secretion decrease, troubles related to breast, babies declining breast and ending breast feeding at an early stage are seen. These problems are related to the self-effıcacy that maternal feels towards breast feeding. The researches show that in addition to the maternal, father's attitude throughout pregnancy is also effective on starting breast feeding, sustaining and maintaining it efficiently.

With this research it has been aimed to evaluate the effect of individual and group breast feeding training of future mother and father at postpartum period on breast-feeding self-effıcacy and attitude.

Research data has been gathered at Turkey Public Hospitals Institution Izmir North Public Hospitals Association of T.R Ministry of Health Tepecik Education and Reserach Hospital between the dates 01 March-30 September 2014.

As a result; it has been seen that breast feeding training is not alone enough to improve self sufficiency and attitude, and maternals have to be supported by health staff at postpartum period in hospital. It is suggested to include also fathers to the breast feeding training provided at pregnancy period.

DETAILED DESCRIPTION:
Breastfeeding training was given to the mother and father candidates in the individual and group education group. At this stage, standard care and service in the hospital was offered to the mothers and fathers in the control group. A follow-up plan was prepared for all the mothers and fathers after the discharge from the phone.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* Having the first pregnancy
* Communicable
* Living with his wife
* Participation in education with his wife
* Completion of 36 weeks of gestational week
* Pregnant women without risk.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Follow-up after discharge | Four months
  Questionnaires were prepared separately for parents in each follow-up. Breastfeeding status, nipple cracking, breastfeeding support status were evaluated in the first week, sixth week and fourth month in the mother follow-up forms.
  The questionnaire to be applied during pregnancy consists of three topics and a total of 25 questions.
  There are questions about the sociodemographic characteristics (10), fertility characteristics (9) and breastfeeding characteristics (6) of the mothers.
  In the questionnaire to be applied in the first week after birth, there are questions about the characteristics of birth and breastfeeding (30).
  In the sixth week, there is a questionnaire (18) containing questions about breastfeeding and finally a questionnaire containing questions about breastfeeding status (18) at the fourth month.
  During the first week, sixth week and fourth month follow-up, fathers' breastfeeding support status was questioned.
Breastfeeding Self-Efficacy Scale: | Four months
  This scale was developed by Cindy-Lee Dennis to measure breastfeeding self-efficacy and consists of 2 sub-scales and 33 items. The cronbach alpha value of the scale developed by Cindy-Lee Dennis was measured as 0.95. The validity and reliability of the breastfeeding self-efficacy scale in Turkish was made by Eksioglu. The Cronbach's alpha coefficient was 0.91 and the Cronbach's alpha coefficient of the "Technical" sub-dimension was 0.89. Breastfeeding self-efficacy increases as the total score increases.The lowest score is 33 and the highest score is 165. The scale was administered to mothers four times. The first application was performed before the training in antenatal period and the other applications were done in the first week, sixth week and fourth month.
IOWA Infant Feeding and Attitude Scale (IIFAS) | Four months
  Developed by De La Mora and Russell, the IIFAS was developed to assess the attitudes of mothers to breastfeeding and consists of 17 items. The cronbach's alpha value of the scale was 0.86. The validity and reliability study in our country was conducted by Eksioğlu et al. And the Cronbach's alpha coefficient was calculated as 0.71. It is designed to estimate the time of breastfeeding as well as choice of infant feeding method.
  Scale; It consists of 17 items evaluated with a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  Nine of the items showed positive formula feeding, whereas these items were counter-rated.
  The total score was between 17 and 85, and the higher the mean score of the scale, the higher the positive attitude of breastfeeding, and the lower the mean score of the scale, the higher the tendency towards formula feeding.
  The scale was applied to the parents four times.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Eidelman AI. Breastfeeding and the use of human milk: an analysis of the American Academy of Pediatrics 2012 Breastfeeding Policy Statement. Breastfeed Med. 2012 Oct;7(5):323-4. doi: 10.1089/bfm.2012.0067. Epub 2012 Sep 4. No abstract available. PMID 22946888
- [Background] Abbass-Dick J, Stern SB, Nelson LE, Watson W, Dennis CL. Coparenting breastfeeding support and exclusive breastfeeding: a randomized controlled trial. Pediatrics. 2015 Jan;135(1):102-10. doi: 10.1542/peds.2014-1416. Epub 2014 Dec 1. PMID 25452653
- [Background] Mangrio E, Persson K, Bramhagen AC. Sociodemographic, physical, mental and social factors in the cessation of breastfeeding before 6 months: a systematic review. Scand J Caring Sci. 2018 Jun;32(2):451-465. doi: 10.1111/scs.12489. Epub 2017 Jun 1. PMID 28569436
- [Background] Maycock B, Binns CW, Dhaliwal S, Tohotoa J, Hauck Y, Burns S, Howat P. Education and support for fathers improves breastfeeding rates: a randomized controlled trial. J Hum Lact. 2013 Nov;29(4):484-90. doi: 10.1177/0890334413484387. Epub 2013 Apr 19. PMID 23603573